CLINICAL TRIAL: NCT03378895
Title: CEPPPIA Pilot. Experimental Center of Participative and Individualized Predictive Prevention in Auvergne
Acronym: CEPPPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: European Regional Development Fund (Other); Conseil Régional Auvergne-Rhône-Alpes, Clermont-Ferrand, France. (Unknown); Agence Régionale de Santé Rhône-Alpes (Other); Ligue Contre le Cancer, Puy de Dôme, Allier et Cantal (Unknown); GIE Auvergne Thermale (Other); Centre Jean Perrin (Other); UFR Médecine (Unknown); UFR STAPS (Unknown); Laboratoire d'Informatique, de Modélisation et d'Optimisation des Systèmes (LIMOS) (Unknown); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-358; 2017-A00666-47 (Other: 2017-A00666-47)
Record Dates: First submitted 2017-10-17; First posted 2017-12-20 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Chronic Disease; Cardiovascular Diseases; Cancers; Diabetes Mellitus; Obesity
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases; Neoplasms; Diabetes Mellitus; Obesity

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults aged 35 to 55 years (Experimental)
  Interventions: Behavioral: online questionnaire

INTERVENTIONS:
Behavioral: online questionnaire — Risk assessment identified by online questionnaire

SUMMARY:
The state of health in France appears to be good with regard to major indicators such as life expectancy at birth.

However, France is characterized by a high standardized rate of premature mortality (deaths occurring before the age of 65) in comparison with other European countries, with geographical disparities. Between 2006 and 2010, the standardized rate of premature mortality was higher in Auvergne than the national average.

Chronic diseases such as cardiovascular diseases, cancers and / or metabolic diseases (including diabetes and obesity) are the main causes of these premature deaths. These diseases have several causes: they depend on the genetic heritage, the way of life and the environment. Family history is a known risk factor for these chronic diseases. Eating habits, insufficient physical activity or physical inactivity, excessive drinking and smoking which promote the occurrence of these chronic diseases are the main risk factors that we can modify. Preventive measures are known and are regularly the subject of public health plans and awareness campaigns targeting lifestyles modification of the populations. These prevention campaigns affect entire population, while the risk factors for chronic diseases are different from one to another, this encourages personalization of preventive measures. The CEPPPIA pilot study falls within this framework and aims to evaluate the feasibility of setting up an individualized prevention program on the modification of health behaviors among people aged 35 to 55, who has a moderate risk of developing chronic diseases and residing in Auvergne territory.

DETAILED DESCRIPTION:
The state of health in France appears to be good with regard to major indicators such as life expectancy at birth.

However, France is characterized by a high standardized rate of premature mortality (deaths occurring before the age of 65) in comparison with other European countries, with geographical disparities. Between 2006 and 2010, the standardized rate of premature mortality was higher in Auvergne than the national average.

Chronic diseases such as cardiovascular diseases, cancers and / or metabolic diseases (including diabetes and obesity) are the main causes of these premature deaths. These diseases have several causes: they depend on the genetic heritage, the way of life and the environment. Family history is a known risk factor for these chronic diseases. Eating habits, insufficient physical activity or physical inactivity, excessive drinking and smoking which promote the occurrence of these chronic diseases are the main risk factors that we can modify. Preventive measures are known and are regularly the subject of public health plans and awareness campaigns targeting lifestyles modification of the populations. These prevention campaigns affect entire population, while the risk factors for chronic diseases are different from one to another, this encourages personalization of preventive measures. The CEPPPIA pilot study falls within this framework and aims to evaluate the feasibility of setting up an individualized prevention program on the modification of health behaviors among people aged 35 to 55, who has a moderate risk of developing chronic diseases and residing in Auvergne territory.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 35 to 55 years
* Subjects identified as moderate risk (group G1) following the assessment of the level of risk
* Covered by the Social Security
* Having signed the information form and having given his / her free consent during the inclusion visit
* Judged able to understand the aims of the study and ready to accept the constraints

Exclusion Criteria:

* Age <35 years or> 55 years
* Person who has not completed and validated the FSI (online health questionnaire)
* Person belonging to group G1 but with a moderate pathological risk (P1) and no identifiable risk in the behavioral field (C0)
* Pregnant or lactating women
* Persons benefiting from a legal protection measure
* Persons refusing to sign information and consent form
* Person in an exclusion period from another study, or having received more than 4500 € in the year
* Person deprived of his liberty by judicial or administrative decision
* Medical or surgical history, judged by the investigator to be incompatible with the study
* Suspicion of psychiatric disorders judged by the investigator to be incompatible with the study

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Individualized Prevention Program participation rate | at day 1
  Number of volunteers who accepted to participate in the interventional phase / number of volunteers who can be included in the study Assess the feasibility of implementing an Individualized Prevention Program on the modification of health behaviors among people aged 35 to 55 years with a risk of developing chronic diseases (cardiovascular diseases, metabolic diseases and / or cancers) and residing in the territory of Auvergne by measuring partipation rate and satisfaction

SECONDARY OUTCOMES:
Variation of the risk score in at least one of the three behavioral domains | at day 1
  Evaluation of the effectiveness of an individualized primary prevention program on changing health behaviors among people aged 35 to 55 years with a risk of developing chronic diseases (cardiovascular diseases, metabolic diseases and/or cancers)
Variation of the risk score in at least one of the three behavioral domains; The risk score will be calculated from the results reported on a self-administered questionnaire | at 3 month
  Evaluate the effectiveness of an individualized primary prevention program on the modification of health behaviors among people aged 35 to 55, at risk of developing chronic diseases (cardiovascular diseases, metabolic diseases and / or cancers) and residing in Auvergne.

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France